CLINICAL TRIAL: NCT04319575
Title: Clinical and Radiographic Comparative Evaluation of Healing of Periapical Lesion Using Triple Antibiotic Paste With Combination of Chitosan and Calcium Hydroxide When Used as a Root Canal Disinfectant- An In Vivo Study
Brief Title: Comparison of Triple Antibiotic Paste With Combination of Chitosan and Calcium Hydroxide as a Root Canal Disinfectant
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, Soumya Shetty, professor, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DYPV/EC/55/16
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Periapical Abscess
MeSH Terms: conditions — Periapical Abscess

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chitosan calcium hyroxide paste (Experimental): after the access preparation and cleaning and shaping, chitosan calcium hydroxide paste will be placed in the canal and kept for 4 weeks.
  Interventions: Drug: root canal treatment and intracanal medicament
- triple antibiotic paste (Active Comparator): after the access preparation and cleaning and shaping, ciprofloxacin metronidazole minocycline paste will be :placed in the canal and kept for 4 weeks.
  Interventions: Drug: root canal treatment and intracanal medicament

INTERVENTIONS:
Drug: root canal treatment and intracanal medicament — after the access preparation and cleaning and shaping was done in 1st appointment using k files,"Mani" and protapers,"Dentsply" then in, chitosan calcium hydroxide paste," or ciprofloxacin metronidazole minocycline paste placed in the canal and kept for 4 weeks.
  Other Names: intra-oral periapical radiaograph,"kodak"

SUMMARY:
Investigators observed the clinical and radiographic healing of periapical lesion using Chitosan mixed with calcium hydroxide and compared it with triple antibiotic paste when used as intracanal medicament in 3months, 6 months and 12 months.

DETAILED DESCRIPTION:
Aim: To evaluate and compare the healing of periapical lesions using chitosan mixed with calcium hydroxide or Triple Antibiotic Paste at 3,6 and 12 months.

Methodology:

20 adult patients having periapical lesions in single rooted teeth were selected in this study after being assessed using the PAI index. Patients were randomly assigned to: Group - I (n=10) Chitosan with Ca (OH)2 and Group -II (n=10) Triple Antibiotic paste (TAP)

After access opening and cleaning and shaping were done in the first visit, the pertinent intracanal medicaments were placed depending on the patient group. After 4 weeks, on the second visit, the medicament was removed andobturation was done in the asymptomatic teeth. Both clinical and radiographic endodontic evaluation was done at 0, 3, 6 and 12months using the same parameters.

Radiographic evaluation was done using the PAI Index and was compared at 0, 3, 6, and 12 months after treatment, Z Test.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 40 years Periapical lesion (not more than 5mm) radiographically.on single rooted teeth
* Roots with closed apex.
* Systemically healthy patients.

Exclusion Criteria:All patients who respond positive to allergic patch test [triple antibiotic paste] and drugs.

* Teeth with previous endodontic therapy performed.
* Patients with a history of any systemic diseases.
* Pregnant and lactating women.
* Tooth associated with vertical root fracture and coronal perforation.
* Tooth affected with calcific degeneration.
* Presence of external or internal root resorption.
* Blunderbuss apex.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-04-23 (Estimated); Study Completion 2020-08-04 (Estimated)

PRIMARY OUTCOMES:
healing of periapical lesion | change in PAI index from baseline to 3 months, baseline to 6 months and baseline to 12 months
  the periapical status will be assessed by using the periapical index [PAI] using radiographs and scoring was done according to following scoring index as
  1. Normal periapical structures
  2. Small changes in bone structure
  3. Changes in bone structure with some mineral loss
  4. Periodontitis with well-defined radiolucent area
  5. Severe periodontitis with exacerbating features

SECONDARY OUTCOMES:
patient pain perception | 3months, 6months and 12 months
  pain will be assessed using visual analogue (VAS )scale along with any swelling following scale of -10 with 0 score depicts no pain and score 10 depicts severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Piyush D Oswal, MDS, Study Director — Dr. D Y Patil Dental College, Pimpri, Pune
Locations (1):
- Dr DY Patil Dental College And Hospital (DPU), Pune, Maharashtra, India